CLINICAL TRIAL: NCT01735461
Title: Oral Calcium Supplementation, a Strategy to Reduce Kidney Stones in Crohn's Patients Living With a Small Bowel Resection
Brief Title: Calcium Supplements Strategy for Kidney Stones Prevention in Crohn's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H11-02525
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Kidney Calculi; Crohn's Disease
MeSH Terms: conditions — Kidney Calculi; Crohn Disease | interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary supplement (Experimental): Calcium Carbonate
  Interventions: Dietary Supplement: Calcium Carbonate

INTERVENTIONS:
Dietary Supplement: Calcium Carbonate — There is a regimen for dietary supplement intake that will be provided to study participants.
  Other Names: CaCO3

SUMMARY:
Hospitalization for kidney stones in the Inflammatory Bowel Disease (IBD) population is common, particularly among Crohn's patients who had a small bowel resection. This patient population experiences a lifetime occurrence of kidney stone formation as high as 25% accompanied with a high rate of recurrence (the typical rate of stone formation is ~10% in the non IBD population). Giving oral calcium is used to bind oxalate in the intestine in an attempt to reduce the amount of oxalate that is absorbed into the body and to reduce urinary oxalate levels. However, there are no defined guidelines for the optimum dosing of calcium. This study's primary objective is to scientifically define an appropriate range of calcium supplementation that reduce the level of oxalate found in the urine of patients living with inflammatory bowel disease.

DETAILED DESCRIPTION:
The primary objective of this study is to establish optimal oral calcium supplementation in Crohn's patients who have had an ileal bowel resection. This population is at high risk for calcium oxalate kidney stones, a direct consequence of extensive gut malabsorption and enteric hyperoxaluria. The benefit of providing oral calcium in this patient population (as a means to reduce intestinal oxalate absorption) is known, however, there are no appropriate targets for calcium dosing, which is presently performed empirically or not at all. Our goal is to establish simple, safe and practical guidelines for calcium supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. a pathologically confirmed diagnosis of Crohn's disease
2. prior ileal resection with an intact colon (surgery>6 months preceding involvement in study)
3. hyperoxaluria (defined as> 48 mg (>0.5 mmol) per 24 hour urine samples.

   * Patients will not be excluded if they are known kidney stone formers.

Exclusion Criteria:

1. current pregnancy
2. patient's without baseline hyperoxaluria (defined as >48 mg or 0.5mmol per 24 hour urine samples)
3. patients in renal failure assessed by a GFR < 60
4. inability to provide informed consent
5. active cancer
6. hyperparathyroidism
7. hyperphosphatemia
8. <19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Molar ratio of urinary calcium:oxalate in relation to the supersaturation product of calcium oxalate | 7 days
  Molar ratio of urinary calcium:oxalate in relation to the supersaturation product of calcium oxalate will be calculated from the 24-hour urine test.
  The patient will take dietary calcium for 7 days and then we will evaluate their urine chemistry. Additionally, 24-hour urine collections are considered the standard for urinalysis in comparison to spot urine chemistry. The initial data, prior to calcium supplementation, will serve as the control, providing the patient's baseline risk for kidney stone formation.

SECONDARY OUTCOMES:
Optimal level of Ca supplementation for prevention of stones in Crohn's patients | 7 days
  Practical guidelines for physicians managing Crohn's patients will be developed based on the optimal Ca supplement dosages and determine the optimal level of calcium supplementation in each patient, based on urinary parameters from 24-hour urine.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No